CLINICAL TRIAL: NCT03163108
Title: Closed-loop Automatic Oxygen Control (CLAC-4) in Preterm Infants: a Randomized Controlled Trial of a Revised Algorithm
Brief Title: Closed-loop Automatic Oxygen Control (CLAC-4) in Preterm Infants
Acronym: CLAC-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Heinen und Löwenstein GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLAC-4
Record Dates: First submitted 2017-03-30; First posted 2017-05-22 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2017-01

CONDITIONS: Infant Respiratory Distress Syndrome; Ventilator Lung; Newborn
Keywords: controller; hyperoxia; hypoxia; ventilation; cerebral oxygenation
MeSH Terms: conditions — Pulmonary Atelectasis; Bronchopulmonary Dysplasia; Hyperoxia; Hypoxia; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RMC only (No Intervention): routine manual control (RMC) of the fraction of inspired oxygen (FIO2)
- CLAC slow (Active Comparator): routine manual control (RMC) + Closed-loop automatic oxygen control (CLAC) with 180sec WAIT-Interval ("slow" algorithm) of the fraction of inspired oxygen (FIO2)
  Interventions: Device: Closed-loop automatic oxygen control (CLAC) slow in addition to RMC
- CLAC fast (Experimental): routine manual control (RMC) + Closed-loop automatic oxygen control (CLAC) with 30sec WAIT-Interval ("fast" algorithm) of the fraction of inspired oxygen (FIO2)
  Interventions: Device: Closed-loop automatic oxygen control (CLAC) fast in addition to RMC

INTERVENTIONS:
Device: Closed-loop automatic oxygen control (CLAC) fast in addition to RMC — Closed-loop automatic oxygen control is an automated, algorithm based adjustment of the fraction of inspired oxygen in relation to arterial saturation (WAIT-interval 30s).
  Arms: CLAC fast
Device: Closed-loop automatic oxygen control (CLAC) slow in addition to RMC — Closed-loop automatic oxygen control is an automated, algorithm based adjustment of the fraction of inspired oxygen in relation to arterial saturation (WAIT-interval 180s).
  Arms: CLAC slow

SUMMARY:
Two-center, randomised controlled, cross-over clinical trial in preterm infants born at gestational age below 34+1/7 weeks receiving supplemental oxygen and respiratory support (Continous positive airway pressure (CPAP) or Non-invasive Ventilation (NIV) or Invasive Ventilation (IV)). Routine manual control (RMC) of the fraction of inspired oxygen (FiO2) will be tested against RMC supported by closed-loop automatic control (CLAC) with "slow"-algorithm and RMC supported by CLAC with "fast"-algorithm.

The primary hypothesis is, that the use of the "faster" algorithm results in more time within arterial oxygen saturation (SpO2) target range compared to RMC only. The a-priori subordinate hypothesis is, that the faster algorithm is equally effective as the slower algorithm to maintain the SpO2 in the target range.

DETAILED DESCRIPTION:
BACKGROUND AND OBJECTIVE In preterm infants receiving supplemental oxygen, routine manual control (RMC) of the fraction of inspired oxygen (FiO2) is often difficult and time consuming. The investigators developed a system for closed-loop automatic control (CLAC) of the FiO2 and demonstrated its safety and efficacy in a multi-center study. The objective of this study is to test a revised, "faster" algorithm with a shorter WAIT-interval of 30sec (= time between FiO2 changes) against the previously tested algorithm (WAIT of 180sec) and against RMC. The primary hypothesis is, that the application of CLAC with the "faster" algorithm in addition to RMC results in more time within arterial oxygen saturation (SpO2) target range compared to RMC only. The a-priori subordinate hypothesis is, that the faster algorithm is equally effective as the slower algorithm to maintain the SpO2 in the target range.

Further hypotheses for exploratory testing are, that the "fast" algorithm will achieve a higher proportion of time with SpO2 within target range and an improved stability of cerebral oxygenation (measured as rcStO2 and rcFtO2E determined by Near-infrared spectroscopy) compared with the slow algorithm.

STUDY DESIGN The Study is designed as a two-center, randomized controlled, cross-over clinical trial in preterm infants receiving mechanical ventilation or nasal continuous positive airway pressure or non-invasive ventilation and supplemental oxygen (FiO2 above 0.21). Within a twenty-four-hour period the investigators will compare 8 hours of RMC with 8-hour periods of RMC supported by CLAC "slow" algorithm or "fast" algorithm, respectively.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth <34+1/7weeks
* invasive mechanical ventilation OR noninvasive ventilation OR continous positive airway pressure support
* Fraction of inspired oxygen above 0.21 before inclusion
* more than 2 hypoxaemic events (arterial oxygen saturation below 80%) within 8 hours before inclusion
* parental written informed consent

Exclusion Criteria:

* congenital pulmonary anomalies
* diaphragmatic hernia or other diaphragmatic disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Proportion of time with SpO2 within target range | 16 hours
  Comparison of proportion of time with SpO2 within target range if the infant requires supplemental oxygen and time above target range if the infant requires no supplemental oxygen between CLAC-fast and RMC (superiority hypothesis).
Proportion of Time with SpO2 within target range | 16 hours
  Comparison of proportion of time with SpO2 within target range if the infant requires supplemental oxygen and time above target range if the infant requires no supplemental oxygen between CLAC-fast and CLAC-slow (subordinate, non inferiority hypothesis).

SECONDARY OUTCOMES:
Duration of hyperoxaemia | 16 hours
  Time with arterial oxygen saturation above 95% if the infant requires supplemental oxygen (hyperoxaemia).
Duration of hypoxaemia | 16 hours
  Time with arterial oxygen saturation below 80% (hypoxaemia)
Duration of "overshoot" hyperoxaemia | 16 hours
  Comparison of proportion of time with SpO2 higher than 95% after an automated increase of FiO2 between CLAC-fast and CLAC-slow.
Number of "overshoot" hyperoxaemia | 16 hours
  Comparison of number of events with SpO2 higher than 95% after an automated increase of FiO2 between CLAC-fast and CLAC-slow.
Stability of cerebral oxygenation | 24 hours
  "Area under the curve" of cerebral tissue saturation or fraction of tissue oxygen extraction outside of the infants Median +- 5% or outside of the "save" interval of 55-80% rcStO2.

OTHER OUTCOMES:
Staff workload | 24 hours
  number of manual adjustments of inspired oxygen per time

CONTACTS AND LOCATIONS:
Overall Officials: Axel R Franz, MD, Principal Investigator — University Hospital Tuebingen
Locations (2):
- Germany (2):
  - Johannes Gutenberg University Mainz, Mainz
  - University of Tubingen, Tübingen

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data is not intended

REFERENCES:
- [Derived] Schwarz CE, Kidszun A, Bieder NS, Franz AR, Konig J, Mildenberger E, Poets CF, Seyfang A, Urschitz MS. Is faster better? A randomised crossover study comparing algorithms for closed-loop automatic oxygen control. Arch Dis Child Fetal Neonatal Ed. 2020 Jul;105(4):369-374. doi: 10.1136/archdischild-2019-317029. Epub 2019 Sep 16. PMID 31527093